CLINICAL TRIAL: NCT03070210
Title: A Randomized, Controlled Trial of Endoscopic Ultrasound Guided Celiac Plexus Blockade (EUS-CPB) With Standard Plexus Injection vs. Direct Celiac Ganglia Block for Treatment of Pain in Chronic Pancreatitis.
Brief Title: Clinical Trial to Evaluate the Endoscopic Ultrasound Guided Celiac Plexus Block for Treatment of Pain in Chronic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Tyler Stevens, Director of Advanced Endoscopy Fellowship Program, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 16-1543
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Pancreatitis, Chronic; Abdominal Pain
MeSH Terms: conditions — Pancreatitis, Chronic; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-celiac plexus block (EUS-CPB) (Other): This is the standard technique. In this approach, the needle is passed through the body of the stomach adjacent the celiac artery into the retroperitoneal space in 1 or 2 passes. The injectate (bupivacaine or alcohol) is injected and spreads through the retroperitoneal space, effectively "bathing" all the ganglia.
  Interventions: Procedure: EUS-celiac plexus block (EUS-CPB)
- EUS-celiac ganglia block (EUS-CGB) (Active Comparator): This is a more recent technique which has been often used. In this procedure, the needle is inserted under EUS guidance directly into as many ganglia as possible. For celiac ganglia <1cm in diameter, the solution is injected into the central point; for those ≥1 cm, a needle is advanced to the deepest point into the ganglia and solution is injected as the needle is slowly withdrawn. Injections are continued until an echogenic pattern is produced over the entire celiac ganglia.
  Interventions: Procedure: EUS-celiac ganglia block (EUS-CGB)

INTERVENTIONS:
Procedure: EUS-celiac ganglia block (EUS-CGB) — The intervention technique of EUS-CGB is the realization of EUS-guided celiac block with injection of bupivacaine directly into the ganglia for patients with chronic pancreatitis.
  Arms: EUS-celiac ganglia block (EUS-CGB)
Procedure: EUS-celiac plexus block (EUS-CPB) — In the arm of EUS-CPB, the procedure is going to be performed with the standard EUS-guided celiac plexus block with injection of bupivacaine into the retroperitoneal space.
  Arms: EUS-celiac plexus block (EUS-CPB)

SUMMARY:
AIM: To compare pain relief in patients randomly assigned to endoscopic ultrasound-guided celiac ganglia block (EUS-CGB) vs standard endoscopic ultrasound-guided celiac plexus block (EUS-CPB).

METHODS: This is a single-center, double-blind, randomized parallel-group study to assess the efficacy of EUS-CPB vs. EUS-CGB in patients with painful chronic pancreatitis.

DETAILED DESCRIPTION:
Inclusion criteria include: age>18 yrs, ability for informed consent, chronic daily pancreatic-type abdominal pain.

Exclusion criteria include: pregnancy, malignancy, recent acute pancreatitis (within 2 months), elevated INR (>1.5) or low platelet count (<75 cells/mm3), allergy to eggs or "caine" anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic pancreatitis and referred for EUS-guided celiac plexus block with: age>18 yrs, ability for informed consent, chronic daily pancreatic-type abdominal pain.

Exclusion Criteria:

* pregnancy, malignancy, recent acute pancreatitis (within 2 months), elevated INR (>1.5) or low platelet count (<75 cells/mm3), allergy to eggs or "caine" anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Pain relief | 1 week
  The primary endpoint will be pain relief at 1 week after the block, defined as a decrease of 3 or more points in the VAS scale measuring "average pain over past week".

SECONDARY OUTCOMES:
Complete response rate | 1 week
  Decrease in pain to 1 or 0.
Duration of pain relief | up to 2 months
  Duration of pain relief will be assessed during a 2-month follow-up.
Opioid consumption | up to 2 months
  Assess the opioid consumption in up to 2 months after endoscopic therapy.
Adverse effects | in up to 2 months
  Assess the incidence of adverse effects after endoscopic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Stevens, MD, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doi S, Yasuda I, Kawakami H, Hayashi T, Hisai H, Irisawa A, Mukai T, Katanuma A, Kubota K, Ohnishi T, Ryozawa S, Hara K, Itoi T, Hanada K, Yamao K. Endoscopic ultrasound-guided celiac ganglia neurolysis vs. celiac plexus neurolysis: a randomized multicenter trial. Endoscopy. 2013;45(5):362-9. doi: 10.1055/s-0032-1326225. Epub 2013 Apr 24. PMID 23616126
- [Background] Ascunce G, Ribeiro A, Reis I, Rocha-Lima C, Sleeman D, Merchan J, Levi J. EUS visualization and direct celiac ganglia neurolysis predicts better pain relief in patients with pancreatic malignancy (with video). Gastrointest Endosc. 2011 Feb;73(2):267-74. doi: 10.1016/j.gie.2010.10.029. PMID 21295640